CLINICAL TRIAL: NCT02965885
Title: A Phase IA/IB Study Evaluating TAS-116 in Patients With Advanced Solid Tumors
Brief Title: A Study of TAS-116 in Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Taiho Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAS-116-101; 10058010 (Other: Taiho Oncology, Inc.); 2015-005328-24 (EudraCT Number)
Record Dates: First submitted 2016-11-10; First posted 2016-11-17 (Estimated); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Advanced Solid Tumors
Keywords: Phase I; Solid Tumors; Pharmacokinetics; Pharmacodynamics; MTD; TAS116; HSP90 Inhibitor; Neoplasms; HER2 positive MBC; NSCLC EGFR; NSCLC ALK positive
MeSH Terms: conditions — Neoplasms | interventions — TAS-116

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TAS-116 (Experimental)
  Interventions: Drug: TAS-116

INTERVENTIONS:
Drug: TAS-116 — TAS-116 is an oral heat shock protein 90 (HSP90) inhibitor investigated in 3 dosing regimens (QD, QOD, 5 days on 2 days off) in patients with advanced solid tumor and then at one dose schedule in advanced breast and lung cancer.

SUMMARY:
A First-in-Human (FIH) study of TAS-116 in patients with advanced solid tumors was first initiated in Japan in April 2014 and has been ongoing since then. The study consists of a dose escalation phase and a dose expansion phase. Three dosing regimens of TAS-116, once daily (QD), every other day (QOD) and 5 days on/2 days off regimens in 21-day cycles, are being evaluated. This phase I study is also planned to enroll patients with advanced solid tumors in UK to confirm the MTD, safety, tolerability, and pharmacokinetics of TAS-116 in a Western patient population in the dose expansion phase. In addition, patients with HER2+ MBC, NSCLC harboring EGFR mutations or NSCLC harbouring ALK translocations will be further evaluated for safety, tolerability, and efficacy in 3 separate cohorts at recommended dose of TAS-116 on the 5 days on/2 days off regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Male or females with an age ≥ 18 years (≥ 20 years in Japan)
2. Patients with histological- or cytological-confirmed, advanced unresectable breast, gastric, or non-small cell lung cancer, who have progressed on (or not been able to tolerate) standard therapy or for whom no standard anticancer therapy exists.

   a. Part C: Only the following subtype of tumors with the molecular/genetic alterations will be enrolled: HER2 positive MBC Advanced NSCLC, harboring EGFR mutations after progression on osimertinib Advanced NSCLC, harboring ALK translocations after treatment with alectinib or at least 2 ALK inhibitors
3. Has At least one measurable lesion as defined by RECIST criteria
4. Is able to take medications orally (e.g., no feeding tube).
5. Is able to agree to and sign informed consent and to comply with the protocol
6. Has adequate organ function

Exclusion Criteria:

1. Has a serious illness or medical condition(s)
2. Has received treatment with any prescribed treatments within specified time frames prior to study drug administration
3. Significant ophthalmologic abnormality,
4. Impaired cardiac function or clinically significant cardiac disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-07-10 (Actual); Primary Completion 2019-05-03 (Actual); Study Completion 2019-05-03 (Actual)

PRIMARY OUTCOMES:
Number of patients experiencing Dose Limiting Toxicity graded according to CTCAE Version 4.03, observed in the Cycle 1 in order to meet the objective of assessment of the MTD of TAS-116 (Part A) | 21 days in Cycle 1
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] (Parts A, B and C) | Safety monitoring will begin at the informed consent obtained and continue up to 28 days after the last dose of TAS-116 or until new anti-tumor therapy, whichever is earlier.
Objective Response Rate using Response Evaluation Criteria in Solid Tumors 1.1 (RECIST) (Part C) | Up to 2 Years

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) after administration of TAS-116 (Parts A and B) | 21 days in Cycle 1
Area under the plasma drug concentration-time curve (AUC) after administration of TAS-116 (Parts A and B) | 21 days in Cycle 1
Disease Control Rate using RECIST 1.1 (Parts A, B, and C) | Up to last participant completes at least 6 months
Duration of Response (Part C) | Up to last participant completes at least 6 months
Progression Free Survival (Part C) | Up to last participant completes at least 6 months
Overall Survival | Up to last participant completes at least 6 months

CONTACTS AND LOCATIONS:
Locations (12):
- United States (3):
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Greenville Health System, Institute for Translational Oncology Research, Greenville, South Carolina
  - US Oncology - Virginia Cancer Specialists, P.C., Fairfax, Virginia
- Italy (4):
  - Policlinico S.Orsola-Malpighi, U.O. Oncologia Medica, Bologna
  - Azienda Ospedaliero-Universitaria Policlinico-Vittorio Emanuele Oncologia Medica, Catania
  - Istituto Europeo di Oncologia , Sviluppo di Nuovi Farmaci per Terapie Innovative, Milan
  - Regina Elena National Cancer Institute, Roma
- United Kingdom (5):
  - Northern Centre for Cancer Care, Newcastle upon Tyne, England
  - Division of Cancer Studies, Kings College London, London
  - Sarah Cannon Research Institute UK, London
  - The Christie NHS Foundation Trust Institute of Cancer Sciences, University of Manchester, Manchester
  - Royal Marsden, Sutton